CLINICAL TRIAL: NCT02324517
Title: Ex Vivo Laboratory Assays Application for Therapy Tailoring in Patients With Severe Bleeding Disorders, Including Hemophilia With Inhibitors
Brief Title: Ex Vivo Laboratory Assays Application for Therapy Tailoring in Patients With Severe Bleeding Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Gila Kenet MD, Director- Thrombosis Unit, Sheba Medical Center
Other Study IDs: SHEBA-09-7563-GK-CTIL
Record Dates: First submitted 2014-11-30; First posted 2014-12-24 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Severe Hemophilia
Keywords: response to various potential therapies as managed by lab assays
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (10):
- Hemophilia: Patients with Hemophilia A OR B
- inhibitor patients: Hemophilia or FXI def with inhibitors
- anticoagulants: patients under therapy with various anticoagulant drugs
- thrombocytopenia: patients with ITP, chronic thrombocytopenia, chemotherapy induced thrombocytopenia
- platelet function disorders: Glanzmann, Bernard Soulier, antiplatelet therapy
- Fibrinogen disordsers: hyperfibrinogenemia, hypofibrinogenemia, dysfibrinogenemia
- acquired hemophilia: patients with autoimmune Ab's to FVIII
- RBD: FXIII DEF, FV+FVIII DEF, FVII DEF, FV DEF
- THROMBOLYTICS: Patients treated by thrombolytic agents
- Hypercoag: thrombophilias, thrombosis- inc under therapy, acquired high thrombotic risk (eg: cancer)

SUMMARY:
Therapy of patients with severe hemophilia (including hemophilia with inhibitors) and other severe bleeding disorders could be monitored and guided based upon special clotting assays , eg thrombin generation and thromboelastography. In this study blood sampled from patients with bleeding disorders will be evaluated applying ex- vivo spiking assays with various coagulation concentrates to potentially address the feasibility of replacement /bypass agents/ combined therapy for future bleeding episodes. Patients that will be further treated by any regimen potentially suggested (as standard care- not within trial) will be thereafter followed , including repeated lab studies to assess the impact of therapy upon hemostasis.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Validated coagulation disorder

Exclusion Criteria:

* Not consenting to participate
* Multiple coagulopathies and comorbidities

Ages: 6 Months to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with coagulopathies (see brief description)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-03; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Thrombin Generation Parameters pre and post therapy / spiking assays | 1 year from enrollment
  Thrombin Generation Parameters (Peak height, ETP) before and after spiking assays with procoagulant drugs will be compared for each patient separately and within each group of patients diagnosed with similar coagulation disorder.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Mediacl Center, Ramat Gan, Israel